CLINICAL TRIAL: NCT05715320
Title: A Randomized, Double Blind, Parallel-controlled Phase 2 Study to Evaluate the Efficacy and Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: Study of CM310 Injection in Subjects With Moderate-to-Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-101109
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): CM310, subcutaneous
  Interventions: Biological: CM310
- Group B (Experimental): CM310, subcutaneous
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — IL-4Rα monoclonal antibody

SUMMARY:
This study is a multi-center, randomized, double-blind, parallel controlled phase 2 study, aimed at evaluating the efficacy and safety of CM310 in the treatment of patients with moderate-to-severe atopic dermatitis, and observing Pharmacokinetics characteristics, Pharmacodynamics effects and immunogenicity.

DETAILED DESCRIPTION:
This study includes screening, treatment and follow-up periods. 160 subjects will be enrolled to receive CM310.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to understand the study and voluntarily sign a written ICF.
* Age ≥ 18 and ≤ 75 years old, male or female.
* The fertile subjects agreed to take effective contraceptive measures throughout the study period.
* The subjects can communicate well with the investigators and complete the follow-up according to the protocol.

Exclusion Criteria:

* Live vaccine or attenuated live vaccine has been vaccinated or planned to be vaccinated within 12 weeks before randomization.
* He received allergen-specific immunotherapy (desensitization therapy) within 6 months before randomization.
* Major surgery is planned during the study period.
* Previous history of atopic keratoconjunctivitis and corneal involvement.
* Other combined skin diseases that may affect the evaluation of the study.
* Confronting IL-4R α Monoclonal antibody or CM310/placebo drug or ingredient allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving EASI-75 | up to week 12
  Proportion of subjects achieving EASI-75 (≥75% reduction from baseline in Eczema Area and Severity Index score).

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China